CLINICAL TRIAL: NCT03990363
Title: A Phase 2b, Multicentre, Randomised, Double-blind, Placebo-controlled Study of Verinurad and Allopurinol in Patients With Chronic KIdney Disease and Hyperuricaemia
Brief Title: A Study of Verinurad and Allopurinol in Patients With Chronic Kidney Disease and Hyperuricaemia
Acronym: SAPPHIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5495C00002
Record Dates: First submitted 2019-05-30; First posted 2019-06-19 (Actual); Results first posted 2023-03-02 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — verinurad; Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- High Dose (Experimental): High Dose (mg) (verinurad/allopurinol) Step 1 - titration_ 3/100 Step 2 - titration_ 7.5/200 Step 3 - target dose_ 12/300
  Interventions: Drug: Verinurad; Drug: Allopurinol
- Intermediate Dose (Experimental): Intermediate Dose (mg) verinurad/allopurinol Step 1 - titration_ 3/100 Step 2 - titration_ 7.5/200 Step 3 - target dose_ 7.5/300
  Interventions: Drug: Verinurad; Drug: Allopurinol
- Low Dose (Experimental): Low Dose (mg) verinurad/allopurinol Step 1 - titration_3/100 Step 2 - titration_3/200 Step 3 - target dose_3/300. As per Protocol Version 5.0, Patients from 3 mg dose will be switched to 24 mg at Visit 9.
  Interventions: Drug: Verinurad; Drug: Allopurinol
- Allopurinol alone (0/300 mg) (Experimental): Step 1 - titration_0/100 Step 2 - titration_0/200 Step 3 - target dose_0/300
  Interventions: Drug: Allopurinol
- Placebo (0/0 mg) (Placebo Comparator): Placebo (mg) in 3 steps_0/0
  Interventions: Drug: Placebo for Verinurad; Drug: Placebo for Allopurinol

INTERVENTIONS:
Drug: Verinurad — Study treatments will be titrated in 3 steps for target low dose (3 mg), intermediate dose ( 7.5 mg) and High Dose (12 mg) Verinurad.
  As per Protocol Version 5.0, Patients from 3 mg dose will be switched to 24 mg at visit 9
  Arms: High Dose; Intermediate Dose; Low Dose
Drug: Allopurinol — Study treatments will be titrated in 3 steps: Low dose (100 mg), intermediate (200 mg) and High Dose ( 300 mg) Allopurinol
  Arms: Allopurinol alone (0/300 mg); High Dose; Intermediate Dose; Low Dose
Drug: Placebo for Verinurad — Matching Capsule
  Other Names: Placebo
  Arms: Placebo (0/0 mg)
Drug: Placebo for Allopurinol — Matching tablet
  Other Names: Placebo
  Arms: Placebo (0/0 mg)

SUMMARY:
The purpose of this clinical research study is to establish the dose of verinurad combined with allopurinol 300 mg once daily that will elicit the desired response; ie, reduction in urinary albumin to creatinine ratio (UACR) at 6 months.

DETAILED DESCRIPTION:
Evidence shows independent associations between hyperuricaemia and the risk of hypertension, myocardial infarction, chronic kidney disease (CKD), type 2 diabetes, heart failure, and metabolic syndrome, including obesity Furthermore, gout, an inflammatory arthritis caused by deposition of monosodium urate crystals in joints, is associated with an increased risk of all-cause death, as well as cardiovascular (CV) death.

Hyperuricaemia is a prerequisite for development of gout, thus linking high levels of sUA to gout and to poor outcomes. However, the causal relationship between hyperuricaemia / gout and the aforementioned diseases and outcomes remains to be proven.

Uric acid transporter 1 (URAT1) is responsible for reabsorption of uric acid (UA in the proximal tubule. Inhibition of URAT1 results in increased urinary excretion of UA.

Verinurad (RDEA3170) is a novel URAT1 inhibitor in Phase 2 development for chronic kidney disease and heart failure.

Verinurad combined with the xanthine oxidase (XO)inhibitor (XOI) febuxostat or allopurinol has been shown to lower sUA in patients with recurrent gout in Phase 2 studies by up to 80%..

The primary objective of this study is to assess the effects of treatment with verinurad and allopurinol, allopurinol alone, and placebo on UACR at 6 months.

In this study, change in UACR at 6 months of treatment is the primary endpoint for the efficacy evaluation of treatment with the combination of verinurad and allopurinol vs. placebo.

A key secondary objective is evaluation of verinurad plus allopurinol on the reduction in UACR at 12 months.

Further, standard safety parameters such as adverse event (AEs), serious adverse event (SAEs), and laboratory evaluations will be employed to assess the safety profile of the study drugs.

Verinurad, allopurinol and oxypurinol plasma concentrations over time will also be measured.

The study will recruit patients with Chronic Kidney Disease and Hyperuricaemia.

ELIGIBILITY:
Inclusion Criteria:

* The subject has given written informed consent prior to any mandatory study specific procedures, sampling, and analyses, and is able to understand and comply with all study procedures
* Adult Patient ≥18 years of age with CKD for >3 months.
* Patients with background standard of care treatment for albuminuria and/or T2DM and treated according to locally recognised guidelines. Therapy optimised and stable for ≥4 weeks before study entry and including an angiotensin-converting enzyme inhibitor or an angiotensin receptor blocker, unless justified.
* If treated with a sodium-glucose transport protein (SGLT2) inhibitor, stable dose for ≥4 weeks before randomisation.
* Meeting screening criteria for sUA and eGFR (Visit 2): sUA ≥6.0 mg/dL. ∙ eGFR ≥25 mL/min/1.73 m2 Chronic Kidney Disease Epidemiology Collaboration
* UACR between 30 mg/g and 5000 mg/g.
* Female patients: Negative pregnancy test for childbearing potential. 1 year post-menopausal, surgically sterile, or using an acceptable method of contraception during the study and 4 weeks after the last dose of study treatment.

Exclusion Criteria:

* Autosomal dominant or autosomal recessive polycystic kidney disease, lupus nephritis or anti-neutrophil cytoplasmic antibody associated vasculitis (granulomatosis with polyangiitis [Wegener's granulomatosis], microscopic polyangiitis, or eosinophilic granulomatosis with polyangiitis [Churg-Strauss syndrome]).
* History of renal transplantation
* Known carrier of the Human Leukocyte Antigen-B *58:01 allele.
* Patients diagnosed with tumor lysis syndrome or Lesch-Nyhan syndrome
* Patients who in the opinion of investigator are unable to perform the patients' tasks associated with the protocol or Presence of any condition which, places the patient at undue risk or potentially jeopardises the quality of the data to be generated
* History of stroke, myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft in the past 6 months
* Uncontrolled hypertension presenting with systolic blood pressure >180 mm Hg and/or diastolic blood pressure >100 mm Hg
* Diagnosed with heart failure and New York Heart Association Functional Classification Class IV at the time of randomisation
* QT interval corrected by the Fridericia formula >470 msec; patients diagnosed with long QT syndrome; patients with a family history of long QT syndrome.
* Subjects with severe hepatic impairment, as judged by the investigator, of Child-Pugh Class C (decompensated cirrhosis), or with major cirrhosis complications (eg, hepatorenal syndrome)
* Receiving cytotoxic or immunosuppressive therapy or other immunotherapy for primary or secondary renal disease within 6 months prior to enrolment
* Treated with any drug for hyperuricaemia in the 6 months preceding randomisation.
* Dose of ACEi, ARBs, fenofibrate, guaifenesin, or SGLT2 inhibitors changed within 4 weeks of randomisation or further dose titration expected after randomization

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 861 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2021-11-22 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (138):
- United States (48):
  - Research Site, Huntsville, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Canyon Country, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Northridge, California
  - Research Site, Orange, California
  - Research Site, Thousand Oaks, California
  - Research Site, Vacaville, California
  - Research Site, Victorville, California
  - Research Site, Denver, Colorado
  - Research Site, Bloomfield, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Altamonte Springs, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Ocala, Florida
  - Research Site, Ocoee, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Wauconda, Illinois
  - Research Site, Paducah, Kentucky
  - Research Site, Takoma Park, Maryland
  - Research Site, Flint, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Jamaica, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Rocky Mount, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Lampasas, Texas
  - Research Site, Lewisville, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Milwaukee, Wisconsin
- Czechia (4):
  - Research Site, Frýdek-Místek
  - Research Site, Prague
  - Research Site, Slaný
  - Research Site, Třebíč
- France (6):
  - Research Site, Annonay
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Rouen
  - Research Site, Tours
- Hungary (9):
  - Research Site, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Hatvan
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Szeged
  - Research Site, Zalaegerszeg
- Israel (15):
  - Research Site, Afula
  - Research Site, Ashdod
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Nazareth
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
  - Research Site, Safed
  - Research Site, Tel Aviv
  - Research Site, Tiberias
- Italy (5):
  - Research Site, Genova
  - Research Site, Milan
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Verona
- Mexico (6):
  - Research Site, Ciudad Madero
  - Research Site, Estado de México
  - Research Site, Guadalajara
  - Research Site, México
  - Research Site, Tijuana
  - Research Site, Veracruz
- Poland (7):
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Romania (5):
  - Research Site, Bucharest
  - Research Site, Deva
  - Research Site, Ploieşti
  - Research Site, Satu Mare
  - Research Site, Timișoara
- Slovakia (9):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Hlohovec
  - Research Site, Košice
  - Research Site, Kráľovský Chlmec
  - Research Site, Lučenec
  - Research Site, Púchov
  - Research Site, Rimavská Sobota
  - Research Site, Svidník
- South Africa (11):
  - Research Site, Benoni
  - Research Site, Cape Town
  - Research Site, Durban
  - Research Site, George
  - Research Site, Johannesburg
  - Research Site, Krugersdorp
  - Research Site, KwaDukuza
  - Research Site, Lenasia
  - Research Site, Paarl
  - Research Site, Pretoria
  - Research Site, Worcester
- Spain (13):
  - Research Site, Alicante
  - Research Site, Barcelona
  - Research Site, Ciudad Real
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, Granada
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Port de Sagunt
  - Research Site, Santander
  - Research Site, Seville
  - Research Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool.
  Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access.
  For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Heerspink HJL, Stack AG, Terkeltaub R, Jongs N, Inker LA, Bjursell M, Maklad N, Perl S, Eklund O, Rikte T, Sjostrom CD, Perkovic V; SAPPHIRE Investigators. Combination Treatment with Verinurad and Allopurinol in CKD: A Randomized Placebo and Active Controlled Trial. J Am Soc Nephrol. 2024 May 1;35(5):594-606. doi: 10.1681/ASN.0000000000000326. Epub 2024 Feb 20. PMID 38564654
- [Derived] Heerspink HJL, Stack AG, Terkeltaub R, Greene TA, Inker LA, Bjursell M, Perl S, Rikte T, Erlandsson F, Perkovic V. Rationale, design, demographics and baseline characteristics of the randomized, controlled, Phase 2b SAPPHIRE study of verinurad plus allopurinol in patients with chronic kidney disease and hyperuricaemia. Nephrol Dial Transplant. 2022 Jul 26;37(8):1461-1471. doi: 10.1093/ndt/gfab237. PMID 34383954
- See also: CSR — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5495C00002&attachmentIdentifier=40101669-5639-49e4-88e0-31ed4e294c1d&fileName=d5495c00002StudySynopsisRedacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled if:
  * serum uric acid was greated than or equal to 6 mg/dL and
  * estimated glomerular filtration rate was greated than or equal to 25 mL/min/1.73 m2 and
  * urinary albumin to creatinine ratio was greated than or equal to 30 mg/g and less than or equal to 5000 mg/g
Groups:
- High Dose: Verinurad 12 mg plus allopurinol 300 mg
- Intermediate Dose: Intermediate dose (verinurad 7.5 mg plus allopurinol 300 mg)
- Low Dose: Verinurad 3 mg plus allopurinol 300 mg.
  As per Protocol Version 5.0, participants from 3 mg dose were switched to 24 mg at Visit 9.
- Allopurinol: Allopurinol alone (Allopurinol): 300 mg
- Placebo: Placebo only
Period: Overall Study
Arm/Group | High Dose | Intermediate Dose | Low Dose | Allopurinol | Placebo
Started | 172 | 172 | 173 | 171 | 173
Switch Dose (As per Protocol Version 5.0, 37 participants from 3 mg dose (ie, Low Dose group) were switched to 24 mg at Visit 9. Participants received Verinurad 24 mg and Allopurinol 300 mg.) | 0 | 0 | 37 | 0 | 0
Completed | 137 | 143 | 131 | 145 | 147
Not Completed | 35 | 29 | 42 | 26 | 26
Not completed — Withdrawal by Subject | 10 | 9 | 18 | 11 | 9
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 2 | 2 | 0
Not completed — Death | 14 | 8 | 14 | 10 | 11
Not completed — Failure to meet randomization criteria | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2
Not completed — Non-compliance with study drug | 2 | 1 | 2 | 0 | 0
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 0 | 0
Not completed — Site terminated by sponsor | 2 | 1 | 2 | 0 | 2
Not completed — Not categorized | 5 | 5 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Inter. Dose: Verinurad 7.5 mg plus allopurinol 300 mg
- Total: Total of all reporting groups
Arm/Group | High Dose | Inter. Dose | Low Dose | Allopurinol | Placebo | Total
Number analyzed (Participants) | 172 | 172 | 173 | 171 | 173 | 861
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at Screening
  Years | 65.3 (10.0) | 64.9 (11.2) | 65.3 (11.2) | 65.1 (11.0) | 65.8 (10.4) | 65.3 (10.8)
Age, Customized [Number; unit: Participants] — Age at Screening
  Participants
    >=65 | 100 | 100 | 107 | 95 | 107 | 509
    <65 | 72 | 72 | 66 | 76 | 66 | 352
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 53 | 57 | 55 | 50 | 284
  Male | 103 | 119 | 116 | 116 | 123 | 577
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 42 | 45 | 37 | 40 | 41 | 205
  Not Hispanic or Latino | 130 | 127 | 136 | 131 | 132 | 656
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — "Unknown or Not Reported" comprises CSR categories "Other" and "Missing".
  Participants
    American Indian or Alaska Native | 4 | 4 | 8 | 5 | 8 | 29
    Asian | 4 | 3 | 5 | 4 | 4 | 20
    Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 0 | 2
    Black or African American | 25 | 24 | 24 | 23 | 20 | 116
    White | 122 | 125 | 126 | 118 | 131 | 622
    More than one race | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 16 | 16 | 10 | 20 | 10 | 72
Region of Enrollment [Count of Participants; unit: Participants] — Country
  Participants
    Czech Republic | 6 | 7 | 3 | 7 | 5 | 28
    France | 2 | 1 | 2 | 0 | 2 | 7
    Hungary | 22 | 25 | 19 | 19 | 22 | 107
    Israel | 15 | 17 | 19 | 15 | 13 | 79
    Italy | 0 | 2 | 0 | 1 | 2 | 5
    Mexico | 6 | 5 | 8 | 7 | 10 | 36
    Poland | 1 | 4 | 2 | 3 | 5 | 15
    Romania | 2 | 5 | 5 | 3 | 7 | 22
    Slovakia | 8 | 6 | 13 | 5 | 6 | 38
    South Africa | 23 | 21 | 20 | 24 | 23 | 111
    Spain | 17 | 12 | 14 | 16 | 17 | 76
    United States | 70 | 67 | 68 | 71 | 61 | 337

OUTCOME MEASURES:

1. Primary Outcome: Urinary Albumin to Creatinine Ratio (uACR) (mg/g) Change From Baseline at 6 Months (Visit 8), Repeated Measures Mixed Model (MMRM)
Description: Analyses of change from baseline in uACR at 6 months (Visit 8) focused on:
  * High dose vs Placebo
  * High dose and Inter. dose combined vs Allopurinol alone
  * Inter. dose vs Placebo
  * Low dose vs Placebo
  * High dose vs Allopurinol
  * Inter. dose vs Allopurinol
  * Low dose vs Allopurinol
  * Allopurinol vs Placebo
  For High dose and Inter. dose combined the 2 categories merged forming 1 new temporary category.
Time Frame: Baseline to 9 months (Visit 9); analysis at 6 months (Visit 8)
Population: Full analysis set (evaluable participant included only)
  In the primary endpoint the arms are presented as comparisons of treatment groups with either placebo or allopurinol alone.
  Geometric mean ratio is presented between arms as a pre-specified analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Groups:
- High Dose Versus Placebo: High dose (verinurad 12 mg plus allopurinol 300 mg) versus placebo
- High Dose and Intermediate Dose Combined Versus Allopurinol: High dose (verinurad 12 mg plus allopurinol 300 mg) and intermediate dose (verinurad 7.5 mg plus allopurinol 300 mg) combined versus allopurinol (allopurinol 300 mg)
- Intermediate Dose Versus Placebo: Intermediate dose (verinurad 7.5 mg plus allopurinol 300 mg) versus placebo
- Low Dose Versus Placebo: Low dose (verinurad 3 mg plus allopurinol 300 mg) versus placebo
- High Dose Versus Allopurinol: High dose (verinurad 12 mg plus allopurinol 300 mg) versus allopurinol (allopurinol 300 mg)
- Intermediate Dose Versus Allopurinol: Intermediate dose (verinurad 7.5 mg plus allopurinol 300 mg) versus allopurinol (allopurinol 300 mg)
- Low Dose Versus Allopurinol: Low dose (verinurad 3 mg plus allopurinol 300 mg) versus allopurinol (allopurinol 300mg)
- Allopurinol Versus Placebo: Allopurinol (allopurinol 300mg) versus placebo
Arm/Group | High Dose Versus Placebo | High Dose and Intermediate Dose Combined Versus Allopurinol | Intermediate Dose Versus Placebo | Low Dose Versus Placebo | High Dose Versus Allopurinol | Intermediate Dose Versus Allopurinol | Low Dose Versus Allopurinol | Allopurinol Versus Placebo
Number analyzed (Participants) | 284 | 434 | 297 | 290 | 283 | 296 | 289 | 291
mg/g | 0.8300 [0.6810 to 1.012] | 1.043 [0.8793 to 1.237] | 0.8369 [0.6887 to 1.017] | 0.8499 [0.6984 to 1.034] | 1.037 [0.8506 to 1.265] | 1.046 [0.8603 to 1.272] | 1.062 [0.8725 to 1.293] | 0.8001 [0.6573 to 0.9739]
Statistical Analysis 1: Comparison: High Dose Versus Placebo; Test type: Superiority; p = 0.0648, Repeated Measures Mixed Model
Statistical Analysis 2: Comparison: High Dose and Intermediate Dose Combined Versus Allopurinol; Test type: Superiority; p = 0.6296, Repeated Measures Mixed Model
Statistical Analysis 3: Comparison: Allopurinol Versus Placebo; Test type: Superiority; p = 0.0263, Repeated Measures Mixed Model

2. Secondary Outcome: Urinary Albumin to Creatinine Ratio (uACR) (mg/g) Change From Baseline at 12 Months (Visit 10), Repeated Measures Mixed Model (MMRM)
Description: Change from baseline in uACR at 12 months (Visit 10) for comparison of Switch dose protocol version 5.0 (PA5) versus double-capsule Placebo.
  The statistical model applied was an MMRM, which was basically the same as the one applied in the primary analysis but adjusted for a 12 month horizon and adapted to the double-capsule regimen from Visit 9 on.
Time Frame: Baseline to 12 months (Visit 10); analysis at 12 months (Visit 10)
Population: Full analysis set (evaluable participant included only)
  In this secondary endpoint the arm presented provides a comparison between the Switch Dose group and double-capsule placebo at Visit 10. This is a pre-specified analysis between the Switch Dose group and double-capsule placebo at Visit 10.
  Geometric mean ratio is presented between arms as a pre-specified analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/g
Groups:
- Switch Dose PA5 Versus Placebo: Switch dose PA5 (verinurad 3 mg plus allopurinol 300 mg up to V9 then verinurad 24 mg plus allopurinol 300 mg) versus placebo
Arm/Group | Switch Dose PA5 Versus Placebo
Number analyzed (Participants) | 78
mg/g | 1.016 [0.7437 to 1.388]

3. Secondary Outcome: Serum Uric Acid (sUA) (mg/dL) Change From Baseline at 6 Months (Visit 8), Repeated Measures Mixed Model (MMRM)
Description: Change from baseline in sUA at 6 months (Visit 8), there were 7 comparisons requested for each endpoint, namely:
  * High dose vs Placebo
  * Inter. dose vs Placebo
  * Low dose vs Placebo
  * High dose vs Allopurinol
  * Inter. dose vs Allopurinol
  * Low dose vs Allopurinol
  * Allopurinol vs Placebo.
Time Frame: Baseline to 9 months (Visit 9); analysis at 6 months (Visit 8)
Population: Full analysis set (evaluable participant included only)
  In this secondary endpoint the arms are presented as comparisons of treatment groups with either placebo or allopurinol alone.
  Geometric mean ratio is presented between arms as a pre-specified analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Groups:
- Interemdiate Dose Versus Allopurinol: Intermediate dose (verinurad 7.5 mg plus allopurinol 300 mg) versus allopurinol (allopurinol 300 mg)
Arm/Group | High Dose Versus Placebo | Intermediate Dose Versus Placebo | Low Dose Versus Placebo | High Dose Versus Allopurinol | Interemdiate Dose Versus Allopurinol | Low Dose Versus Allopurinol | Allopurinol Versus Placebo
Number analyzed (Participants) | 285 | 297 | 291 | 280 | 292 | 286 | 289
mg/dL | 0.5098 [0.4701 to 0.5528] | 0.5810 [0.5362 to 0.6295] | 0.6096 [0.5623 to 0.6609] | 0.8184 [0.7544 to 0.8878] | 0.9327 [0.8604 to 1.011] | 0.9786 [0.9024 to 1.061] | 0.6229 [0.5744 to 0.6755]

4. Secondary Outcome: Serum Uric Acid (sUA) Change From Baseline at 12 Months (Visit 10), Repeated Measures Mixed Model (MMRM)
Description: Change from baseline in sUA at 12 months (Visit 10) for comparison of Switch dose protocol version 5.0 (PA5) versus double-capsule Placebo.
Time Frame: Baseline to 12 months (Visit 10); analysis at 12 months (Visit 10)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Switch Dose PA5 Versus Placebo
Number analyzed (Participants) | 74
mg/dL | 0.5540 [0.4825 to 0.6362]

5. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) (mL/Min/1.73 m²) Change From Baseline at 6 Months (V8), Repeated Measures Mixed Model (MMRM)
Description: Change from baseline in eGFR at 6 months (Visit 8), there were 7 comparisons requested for this endpoint, namely:
  * High dose vs Placebo
  * Inter. dose vs Placebo
  * Low dose vs Placebo
  * High dose vs Allopurinol
  * Inter. dose vs Allopurinol
  * Low dose vs Allopurinol
  * Allopurinol vs Placebo.
Time Frame: Baseline to 9 months (Visit 9); analysis at 6 months (Visit 8)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mL/min/1.73 m²
Arm/Group | High Dose Versus Placebo | Intermediate Dose Versus Placebo | Low Dose Versus Placebo | High Dose Versus Allopurinol | Interemdiate Dose Versus Allopurinol | Low Dose Versus Allopurinol | Allopurinol Versus Placebo
Number analyzed (Participants) | 285 | 297 | 291 | 280 | 292 | 286 | 289
mL/min/1.73 m² | 1.009 [0.9647 to 1.056] | 0.9730 [0.9307 to 1.017] | 1.010 [0.9660 to 1.056] | 1.023 [0.9773 to 1.070] | 0.9859 [0.9429 to 1.031] | 1.024 [0.9786 to 1.071] | 0.9868 [0.9436 to 1.032]

6. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR) (mL/Min/1.73 m²) Change From Baseline at 12 Months (Visit 10)
Description: Change from baseline in eGFR at 12 months (Visit 10) for the following treatments:
  * High Dose
  * Inter. Dose
  * Low Dose (a)
  * Switch Dose protocol version 5.0 (PA5) (b)
  * Allopurinol
  * Placebo
    1. Subjects that switched from Verinurad 3 mg to Verinurad 24 mg at Visit 9 are not included in this group for Visit 10.
    2. Contains all subjects randomized to the low dose group that later switched to Verinurad 24 mg plus Allopurinol 300 mg.
Time Frame: Change from baseline to 12 months (Visit 10)
Population: Full analysis set (evaluable participant included only)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/1.73 m²
Groups:
- High Dose: High dose (verinurad 12 mg plus allopurinol 300 mg)
- Low Dose: Low dose (verinurad 3 mg plus allopurinol 300 mg)
- Switch Dose PA5: Switch dose PA5 (verinurad 3 mg plus allopurinol 300 mg up to V9 then verinurad 24 mg plus allopurinol 300 mg)
- Allopurinol: Allopurinol (allopurinol 300 mg)
Arm/Group | High Dose | Intermediate Dose | Low Dose | Switch Dose PA5 | Allopurinol | Placebo
Number analyzed (Participants) | 124 | 137 | 99 | 34 | 131 | 138
mL/min/1.73 m² | 0.9809 (20.09) | 0.9454 (21.24) | 0.9613 (17.59) | 1.101 (27.23) | 0.9593 (23.36) | 0.9469 (23.33)

7. Secondary Outcome: S-creatinine (mg/dL) Change From Baseline at 6 Months (V8), Repeated Measures Mixed Model (MMRM)
Description: Change from baseline in S-creatinine at 6 months (Visit 8), there were 7 comparisons requested for this endpoint, namely:
  * High dose vs Placebo
  * Inter. dose vs Placebo
  * Low dose vs Placebo
  * High dose vs Allopurinol
  * Inter. dose vs Allopurinol
  * Low dose vs Allopurinol
  * Allopurinol vs Placebo.
Time Frame: Baseline to 9 months (Visit 9); analysis at 6 months (Visit 8)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Ratio
Arm/Group | High Dose Versus Placebo | Intermediate Dose Versus Placebo | Low Dose Versus Placebo | High Dose Versus Allopurinol | Interemdiate Dose Versus Allopurinol | Low Dose Versus Allopurinol | Allopurinol Versus Placebo
Number analyzed (Participants) | 285 | 297 | 291 | 280 | 292 | 286 | 289
Geometric Mean Ratio | 0.9888 [0.9523 to 1.027] | 1.023 [0.9857 to 1.062] | 0.9901 [0.9538 to 1.028] | 0.9801 [0.9437 to 1.018] | 1.014 [0.9770 to 1.053] | 0.9814 [0.9452 to 1.019] | 1.009 [0.9718 to 1.047]

8. Secondary Outcome: S-creatinine (mg/dL) Change From Baseline at 12 Months (Visit 10)
Description: Change from baseline in S-creatinine at 12 months (Visit 10) for the following treatments:
  * High Dose
  * Inter. Dose
  * Low Dose (a)
  * Switch Dose protocol version 5.0 (PA5) (b)
  * Allopurinol
  * Placebo
    1. Subjects that switched from Verinurad 3 mg to Verinurad 24 mg at Visit 9 are not included in this group for Visit 10.
    2. Contains all subjects randomized to the low dose group that later switched to Verinurad 24 mg plus Allopurinol 300 mg.
Time Frame: Change from baseline to 12 months (Visit 10)
Population: Full analysis set (evaluable participant included only)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/dL
Arm/Group | High Dose | Intermediate Dose | Low Dose | Switch Dose PA5 | Allopurinol | Placebo
Number analyzed (Participants) | 124 | 137 | 99 | 34 | 131 | 138
mg/dL | 1.011 (18.57) | 1.038 (18.37) | 1.026 (17.15) | 0.9078 (17.66) | 1.028 (24.44) | 1.043 (20.91)

9. Secondary Outcome: P-cystatin C (mg/L) Change From Baseline at 6 Months (V8), Repeated Measures Mixed Model (MMRM)
Description: Change from baseline in P-cystatin C at 6 months (Visit 8), there were 7 comparisons requested for this endpoint, namely:
  * High dose vs Placebo
  * Inter. dose vs Placebo
  * Low dose vs Placebo
  * High dose vs Allopurinol
  * Inter. dose vs Allopurinol
  * Low dose vs Allopurinol
  * Allopurinol vs Placebo.
Time Frame: Baseline to 9 months (Visit 9); analysis at 6 months (Visit 8)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Ratio
Arm/Group | High Dose Versus Placebo | Intermediate Dose Versus Placebo | Low Dose Versus Placebo | High Dose Versus Allopurinol | Interemdiate Dose Versus Allopurinol | Low Dose Versus Allopurinol | Allopurinol Versus Placebo
Number analyzed (Participants) | 288 | 299 | 294 | 281 | 292 | 287 | 291
Geometric Mean Ratio | 1.009 [0.9758 to 1.042] | 1.038 [1.005 to 1.073] | 1.018 [0.9856 to 1.052] | 0.9849 [0.9528 to 1.018] | 1.014 [0.9813 to 1.048] | 0.9946 [0.9623 to 1.028] | 1.024 [0.9908 to 1.058]

10. Secondary Outcome: P-cystatin C (mg/L) Change From Baseline at 12 Months (Visit 10)
Description: as for outcome 8
Time Frame: Change from baseline to 12 months (Visit 10)
Population: Full analysis set (evaluable participant included only)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | High Dose | Intermediate Dose | Low Dose | Switch Dose PA5 | Allopurinol | Placebo
Number analyzed (Participants) | 124 | 141 | 99 | 34 | 131 | 138
mg/L | 1.070 (17.98) | 1.079 (15.63) | 1.065 (16.51) | 1.018 (13.68) | 1.083 (23.13) | 1.048 (14.89)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Visit 3 (Week 0) until End of Treatment Visit, Visit 10 (Week 60).
Description: From Visit 3 until Visit 10, instances of death, serious adverse events, and non-serious adverse events (with a frequency of >5%) are presented.
  The exposure was shorter in the Low Dose and Switch Dose arms, since this is while under 3 mg treatment up to Visit 10 or beyond and while under 24 mg treatment from Visit 9 to Visit 10, respectively.
  There were 14 subjects that started on Low Dose that died, 1 of these died during the period in which they had changed to the Switch Dose group.
Groups:
- Switch Dose: As per Protocol Version 5.0, participants from 3 mg dose (ie, Low Dose group) were switched to 24 mg at Visit 9. Participants received Verinurad 24 mg and Allopurinol 300 mg.
Arm/Group | High Dose | Intermediate Dose | Low Dose | Switch Dose | Allopurinol | Placebo
All-Cause Mortality (participants affected / at risk) | 14/172 | 8/172 | 13/172 | 1/37 | 10/171 | 11/173
Serious Adverse Events (participants affected / at risk) | 36/172 | 39/172 | 40/172 | 4/37 | 42/171 | 35/173
Other Adverse Events (participants affected / at risk) | 32/172 | 32/172 | 28/172 | 1/37 | 39/171 | 49/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=172) | Intermediate Dose (N=172) | Low Dose (N=172) | Switch Dose (N=37) | Allopurinol (N=171) | Placebo (N=173)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to the mediastinum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (5)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paroxysmal atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Death (General disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 6 (6) | 4 (4)
Covid-19 pneumonia (Infections and infestations) | 4 (4) | 3 (3) | 5 (5) | 0 (0) | 3 (3) | 3 (3)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sars-cov-2 test positive (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Dose (N=172) | Intermediate Dose (N=172) | Low Dose (N=172) | Switch Dose (N=37) | Allopurinol (N=171) | Placebo (N=173)
Headache (Nervous system disorders) | 8 (9) | 4 (4) | 6 (6) | 0 (0) | 3 (4) | 11 (13)
Hypertension (Vascular disorders) | 6 (6) | 9 (12) | 5 (7) | 0 (0) | 12 (13) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 5 (5) | 2 (2) | 1 (1) | 8 (9) | 11 (12)
Blood creatinine increased (Investigations) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 9 (10) | 2 (8)
Gout (Metabolism and nutrition disorders) | 3 (3) | 6 (7) | 9 (9) | 0 (0) | 5 (7) | 13 (19)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (4) | 3 (3) | 0 (0) | 5 (5) | 10 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (10) | 5 (6) | 4 (4) | 1 (1) | 5 (6) | 11 (11)

LIMITATIONS AND CAVEATS:
The study was initially planned to be 108 weeks. However, following the implementation of the amendment in Protocol Version 5.0, all patients discontinued therapy after 60 weeks (Visit 10).

Subjects that were on Low dose at Visit 9 were switched to 24 mg dose.

The study was terminated in Mexico in March 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03990363/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT03990363/SAP_001.pdf